CLINICAL TRIAL: NCT02098928
Title: Multicenter Randomized Controlled Trial on Comparison of Efficacy Between Hand Acupuncture and Electro-acupuncture in Treatment of Menopausal Hot Flashes Symptoms
Brief Title: Comparison Between Hand-acupuncture and Electro-acupuncture Stimulation in the Treatment of Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Collaborators: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012BAI24B01
Record Dates: First submitted 2014-03-05; First posted 2014-03-28 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2014-03

CONDITIONS: Menopause; Puncture Site Reaction
Keywords: Acupuncture; Electro acupuncture; Menopause

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hand-acupuncture group (Active Comparator): Use Hand-acupuncture directly. Four acupoints:Tianshu,Zigong,Guanyuan and Sanyinjiao. Every patient are supposed to have 24 times acupuncture treatment. 30 minutes per time.
  Interventions: Behavioral: Hand-acupuncture; Device: Electrico-acupuncture
- Electric-acupuncture group (Placebo Comparator): Use Electrico-acupuncture device to therapy. Four acupoints:Tianshu,Zigong,Guanyuan and Sanyinjiao. Every patient are supposed to have 24 times acupuncture treatment. 30 minutes per time.
  Interventions: Behavioral: Hand-acupuncture; Device: Electrico-acupuncture

INTERVENTIONS:
Behavioral: Hand-acupuncture — Use Hand-acupuncture directly. Four acupoints:Tianshu,Zigong,Guanyuan and Sanyinjiao. Every patient are supposed to have 24 times acupuncture treatment. 30 minutes per time.
  Other Names: Use Hua Tuo brand disposable acupuncture needles
Device: Electrico-acupuncture — Use Electrico-acupuncture device to therapy. Four acupoints:Tianshu,Zigong,Guanyuan and Sanyinjiao. Every patient are supposed to have 24 times acupuncture treatment. 30 minutes per time.
  Other Names: SDZ electro-acupuncture device

SUMMARY:
Main objective: to compare the effects of hand-acupuncture and electro-acupuncture stimulation on the baking heat symptoms of menopause Secondary objective: to evaluate the safety and acceptability of hand acupuncture and electroacupuncture stimulation

ELIGIBILITY:
Inclusion Criteria:

1. in past of 12 months in, menstrual cycle not rules, menstrual ahead of or wrong Hou ≥ 7 days (menopause transition period early); in past of 12 months in, at least shedding had 2 a menstrual cycle, or amenorrhea over 60 days, but ≤ November (menopause transition period late); last once menstrual to stopped by Hou 3 years within (menopause 3 years within patients)
2. Menopause-related symptoms: baking heat, sweating, insomnia, migraines,irritability, sore vagina, sexual intercourse and so on
3. 40-55 years
4. Baseline scorch score ≥ 6 points
5. without hormone therapy indications for mandatory, such as during menopause, osteoporosis mobility
6. volunteered for this study, and sign the consent form

Exclusion Criteria:

1. test within 3 months before the menstrual cycle rules
2. nearly 4 weeks applied estrogen, SSRIs, soy isoflavones, progesterone, vitamin e, or Black Cohosh
3. diameter greater than 4cm fibroid ovarian cyst, ovarian or after hysterectomy
4. disease history of chemotherapy or who are undergoing chemotherapy
5. unexplained vaginal bleeding
6. coagulation disorders or taking anticoagulant drugs such as warfarin, heparin
7. suffered from skin diseases like eczema, psoriasis, etc
8. severe hepatic and renal insufficiency
9. yet controlled high blood pressure, diabetes, or thyroid disease
10. diabetic nerve damage, cancer and mental illnesses (including depression)
11. wishes are in pregnancy or pregnancy or breastfeeding
12. long-term use of sedatives or antidepressants
13. long-term smoking and alcoholism
14. installed pacemaker or artificial joints

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in average scores of 24-hour hot flashes symptoms at 32 weeks | into the group, into the group after the 4th, 8, 20 and 32 weeks.
  The average scores of 24 hours hot flashes integration consists of integrating the hot flashes times and hot flashes extent, hot flashes degree of mild, moderate and severe hot flashes three categories. Recorded by diary cards of hot flashes symptoms diary cards.

SECONDARY OUTCOMES:
Scores of menopause rating scale（MRS） | into the group, into the group after the 4th, 8, 20 and 32 weeks.
Scores of Menopause-Specific Quality of Life Questionnaire （MENQOL） | into the group, into the group after the 4th, 8, 20 and 32 weeks.
Scores of the Self-Rating Anxiety Scale（SAS） | into the group, into the group after the 4th, 8, 20 and 32 weeks.
Scores of the Self-rating depression scale（SDS） | into the group, into the group after the 4th, 8, 20 and 32 weeks.
the serum levels of sex hormones | into the group, into the group after the 8th week; secondary evaluation points: into the group after the 20th week.
  Menstruation are required in the first 2-4 days of the menstrual blood test, then if no menstruation, menstrual cycles can wait until next month before testing; menopause, while those in the first eight weeks and 20 weekend testing.

OTHER OUTCOMES:
safety evaluation of acupuncture | immediate records
  Content including broken needle, and left needle, and during, and acupuncture pain and the VAS scoring, and difficult endured of acupuncture pain (VAS ≥ 8 points, 10 points system), and needle Hou pain and the scoring, and continued time over 2 hours of more dramatic of needle Hou pain (VAS ≥ 4 points, 10 points system), and local hematoma, and infection or abscess; acupuncture Hou other does not apply sense (refers to acupuncture Hou appeared of fatigue, and palpitations, and dizzy, and headache, and insomnia, symptoms of VAS scoring of average degree and the average continued time; other is not foreseen of bad event. Form sheet for specific, when the diagnosis and treatment of patients at a time, asks if there are adverse events and reactions, if any, immediate records.
evaluation of discomfort when acupuncturing | 1TH and 12th within 5 minutes after the end of acupuncture treatment, take these two averages. Where a VAS value is missing, a VAS for the result.
  evaluation of VAS maximum discomfort occurs during treatment.
subjects acceptance evaluation | 1TH and 12th at the end of treatment with acupuncture and moxibustion, and taking the average.
  an evaluation using the 0-4 system, that is divided into unacceptable (0 points), is more difficult to accept (1), moderate access (2 points), the more acceptable (3 points), very easy to take (4 points), causes unacceptable to write out.
health economics indexes | into the group after 8th during recording.
  Includes direct medical costs (check fees, fees and other costs of acupuncture and moxibustion) and hidden costs (such as round trip transportation, lost)
research evaluation | to 32nd after into the Group during recording
  Compliance, rejection and expulsion rates

CONTACTS AND LOCATIONS:
Overall Officials: zhang wei, Professor, Study Chair — The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine
Locations (1):
- The first affiliate hospital of Hunan university of chinese traditional medicine, Changsha, Hunan, China